CLINICAL TRIAL: NCT01809093
Title: Modulation of Thrombospondin-1 and Pigment Epithelium Derived Factor Levels in Vitreous Fluid and Plasma of Patients With Diabetes
Brief Title: Thrombospondin-1 and Pigmented Epithelium Derived Factor Levels in Patients With Diabetes Mellitus.
Acronym: PEDF
Status: Completed | Type: Observational
Sponsor: MidAtlantic Retina (Other)
Responsible Party: Sponsor-Investigator, MidAtlantic Retina, Principal Investigator, Wills Eye
Organization: Wills Eye (Other)
Other Study IDs: 09-954; IRB# 09-954 (Other: Wills Eye Health System IRB)
Record Dates: First submitted 2013-03-07; First posted 2013-03-12 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Diabetes; Diabetes Mellitus
Keywords: PEDF; TSP1; Thrombospondin; pigment epithelium derived factor; Wills Eye Institute; Pars plana vitrectomy; Vitreous levels; Mid Atlantic Retina; Blood draw; Blood test
MeSH Terms: conditions — Diabetes Mellitus | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The level of TSP1 and PEDF in the vitreous and plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood draw: Blood (approximately equal to 3 to 4 tablespoons) will be drawn at the Wills Eye Institute, 1 time.
  Interventions: Biological: Blood draw

INTERVENTIONS:
Biological: Blood draw — 3-4 tablespoons of blood will be drawn, one time.

SUMMARY:
You are being asked to be in a research study to determine blood levels and vitreous levels of compounds called thrombospondin 1 (TSP1) and pigment epithelium derived factor (PEDF). These compounds exists naturally in your body.

DETAILED DESCRIPTION:
The hypothesis tested here is that diabetic patients that express the higher molecular weight pigment epithelium-derived factor (PEDF) isoform have lower thrombospondin-1 (TSP1) level and, as a result, are at a greater risk for the development of more severe diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Diabetes Mellitus
* Undergoing pars plana vitrectomy for any reason

Exclusion Criteria:

* Use of any anti-VEGF (vascular endothelial growth factor ) medications

Min Age: 18 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus who are undergoing pars plana vitrectomy for any reason
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2010-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Level of thrombospondin (TSP1) and pigment epithelium derived factor (PEDF) in the vitreous and plasma | up to 6 months
  Your voluntary participation in this study may help determine how different TSP1 and PEDF levels correlate with diabetic eye disease.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Spirn, M.D., Principal Investigator
Locations (1):
- Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No